CLINICAL TRIAL: NCT04765722
Title: Mepolizumab for the Treatment of Chronic Cough With Eosinophilic Airways Diseases
Acronym: MUCOSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISS-21-4463
Record Dates: First submitted 2021-02-05; First posted 2021-02-21 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: Chronic Cough; Eosinophilic Bronchitis; Asthma
Keywords: Mepolizumab; Treatment; Anti-interleukin-5; Proof-of-concept study; Randomized; Double-blind; Placebo controlled
MeSH Terms: conditions — Chronic Cough; Asthma | interventions — mepolizumab; Saline Solution

STUDY DESIGN:
Intervention Model Description: Single-centre, randomized, double-blind, placebo-controlled, parallel-group proof-of-concept study to evaluate the effectiveness of 4 doses of mepolizumab for the treatment of refractory chronic cough in patients with asthma and non-asthmatic eosinophilic bronchitis. The study will have 2 arms, each with 15 participants, and a total of 9 visits per subject. Subjects will be screened and within 2 weeks randomized to the intervention (mepolizumab) or placebo arm. Subjects will receive the intervention over a 12 week period at visits 3, 4, 5, and 7. The primary outcome will be measured at visit 14 which will occur 2 weeks after the final intervention dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be assigned to one of the two possible treatment arms generated by a computer-generated randomization schedule prepared by McMaster University, with a ratio of 1:1, mepolizumab or placebo. As there is a known imbalance in the prevalence and cough rates, the study will include sex as a randomization factor. This will mitigate the possibility of the intervention being confounded by sex differences in the 2 arms of the study. Blinded study drug supplies will be provided in sequentially numbered identical syringes in accordance with the randomization schedule and dispensed by a pharmacist who shall not be delegated any other role in the study. Subjects, investigators, research staff (with the exception of the pharmacist) and the sponsor will be masked to the treatment sequence assignment. A sealed code-break envelope for each subject containing details of the treatment allocated will be kept in a locked safe at the study site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepolizumab arm (Experimental): Mepolizumab Dosage form: 1ml pre-filled syringe Dosage: 100mg Frequency: 4 doses at days 0, 28, 56 and 84 Duration: 12 weeks
  Interventions: Drug: Mepolizumab
- Placebo arm (Placebo Comparator): Normal Saline (0.09% normal saline) Dosage form: 1ml pre-filled syringe Dosage: n/a Frequency: 4 doses at days 0, 28, 56 and 84 Duration: 12 weeks
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab subcutaneous injection administered 4 times days 0, 28, 56 and 84 during 12 week treatment period.
  Other Names: Nucala
  Arms: Mepolizumab arm
Drug: Normal Saline — Placebo subcutaneous injection administered 4 times days 0, 28, 56 and 84 during 12 week treatment period.
  Other Names: 0.09% normal saline
  Arms: Placebo arm

SUMMARY:
Cough is the most common presenting symptom to family physician. Chronic Cough affects approximately 10-12% of the general population and is one of the commonest reasons for referral to secondary care. Unfortunately, there are no licensed treatments for this debilitating condition, which is associated with a poor quality of life, affecting the social, physical and psychological well-being of patients.

The aim of this single-centre proof-of-concept study is to investigate whether mepolizumab reduces objective cough frequency in patients with eosinophilic asthma and non-asthmatic eosinophilic bronchitis presenting with chronic cough. Secondary outcomes including the effects on quality of life, the intensity of irritant sensations, airway hyper-reactivity and inflammatory cells and their progenitors will also be evaluated.

The investigators hypothesize that in patients with asthma and non-asthmatic eosinophilic bronchitis, eosinophils are involved in sensitizing airway nerves and thereby increasing spontaneous objective coughs. The investigators predict that treatment with mepolizumab will reduce airway eosinophilia in patients with chronic cough due to eosinophilic asthma and non-asthmatic eosinophilic bronchitis, thereby causing a reduction in objective cough frequency.

DETAILED DESCRIPTION:
This is a 9-visit randomized, double-blind, placebo-controlled, parallel-group Phase IV study. The purpose of this study is to evaluate the effectiveness of mepolizumab for the treatment of refractory chronic cough in patients with eosinophilic airway disease. Patients will be recruited from secondary care clinics. Patient eligibility will be assessed against the study inclusion/exclusion criteria and patients will undergo informed consent in the research centre. Subjects who provide informed consent and are enrolled in the study will undergo screening procedures.

The study will consist of a Mepolizumab treatment arm and placebo arm (normal saline). Fifteen subjects will be randomly assigned to the treatment arm and fifteen subjects will be randomly assigned to the placebo arm in a 1:1 ratio. Following screening and randomization, subjects will under an 12-week treatment period during which they will receive 4 doses of the study drug at days 0, 28, 56, and 84. The primary study outcomes will be measured at week 14 week, 2 weeks following the treatment period.

At Visit 1 (screening), subjects will undergo screening procedures: complete medical history, physical examination, methacholine challenge, spirometry, sputum induction, and blood sampling. Subjects will complete the Leicester Cough Questionnaire and modified Borg Scale.

At Visit 2, subjects will be fitted with a 24-hour cough monitor.

At Visit 3, 24-hour cough monitors will be removed and subjects will undergo spirometry, blood sampling and sputum induction. Subjects will complete the Leicester Cough Questionnaire, modified Borg Scale, and Cough Severity Visual Analogue Scale. The first dose of the study drug will be administered in the clinical research facility by a study physician.

At Visit 4, subjects will undergo spirometry and blood sampling and complete the Leicester Cough Questionnaire, modified Borg Scale, and Cough Severity Visual Analogue Scale. The second dose of the study drug will be administered in the clinical research facility by a study physician.

At Visit 5, the third dose of the study drug will be administered in the clinical research facility by a study physician. Subjects will be fitted with a 24-hour cough monitor.

At Visit 6, 24-hour cough monitors will be removed and subjects will undergo spirometry, sputum induction and blood sampling and complete the Leicester Cough Questionnaire, modified Borg Scale, and Cough Severity Visual Analogue Scale.

At Visit 7, subjects will undergo spirometry and blood sampling and complete the Leicester Cough Questionnaire, modified Borg Scale, and Cough Severity Visual Analogue Scale. The fourth dose of the study drug will be administered in the clinical research facility by a study physician.

At Visit 8, subjects will be fitted with a 24-hour cough monitor.

At Visit 9, the 24-hour cough monitors will be removed and subjects will undergo spirometry, methacholine challenge, sputum induction, and blood sampling. Subjects will complete the Leicester Cough Questionnaire, modified Borg Scale, and Cough Severity Visual Analogue Scale.

All study procedures will be performed according to local standard operating procedures and be conducted by trained and experienced staff with supervision by medical doctors. Study physicians will administer all study drug injections. Safety will be assessed throughout the study by monitoring for adverse events and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18
2. Subjects with a history of chronic cough (cough lasting for >8 weeks)
3. Evidence of airway eosinophilia (sputum eosinophilia>2%)
4. Forced expiratory volume-1 ≥ 70% of predicted
5. Normal chest x-ray (within the last 6 months)
6. At least one dose of a COVID-19 vaccine a minimum of 2 weeks prior to enrollment

Exclusion Criteria:

1. Symptoms of upper respiratory tract infection in the last 1 month which have not resolved.
2. Lower respiratory tract infection or pneumonia in the last 1 month.
3. Subjects with a positive covid-19 test within 2 weeks of screening
4. Subjects with seasonal allergic rhinitis that affects their asthma control
5. Current smoker or ex-smoker with ≥10 pack year smoking history and abstinence of ≤6 months
6. Symptoms of uncontrolled asthma at screening defined as: Asthma Control Questionnaire-5 >1.5, or use of 3 or more puffs of a short acting beta-2 agonist per week, or an exacerbation in the previous month requiring oral prednisone or antibiotics.
7. Use of regular maintenance oral corticosteroids or long-acting muscarinic antagonist within 4 weeks prior to enrolment into the study.
8. A previous asthma exacerbation requiring Intensive Care Unit admission.
9. Significant other primary pulmonary disorders in particular; pulmonary embolism, pulmonary hypertension, interstitial lung disease, lung cancer, cystic fibrosis, emphysema or bronchiectasis.
10. Any history or symptoms of cardiovascular disease, particularly coronary artery disease, arrhythmias, hypertension, or congestive heart failure.
11. Any history or symptoms of significant neurologic disease, including transient ischemic attack, stroke, seizure disorder, or behavioural disturbances
12. Uncontrolled diabetes
13. End-stage kidney or liver disease
14. Clinically significant abnormalities in laboratory test results during the screening period (including complete blood count, coagulation, electrolytes, liver function tests) unless deemed not significant by the investigator.
15. Any history or symptoms of clinically significant autoimmune disease
16. History of anaphylaxis to any biologic therapy or vaccine
17. History of Guillain-Barre Syndrome
18. A helminth parasitic infection diagnosed within 24 weeks prior to the date of informed consent is obtained that has not been treated with or has failed to respond to standard of care therapy.
19. Positive hepatitis B surface antigen, or hepatitis C virus antibody serology, or a positive medical history for hepatitis B or C. Subjects with a history of hepatitis B vaccination without history of hepatitis B can enroll.
20. A history of immunodeficiency disorders including a positive human immunodeficiency virus test
21. Pregnancy or breast-feeding.
22. Women of childbearing potential must not be actively seeking pregnancy, and must use an effective form of birth control (confirmed by the Investigator). Effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective intrauterine device/ intrauterine system levonorgestrel Intrauterine system, Depo-Provera™ injections, oral contraceptive, and Evra Patch™ or Nuvaring™. Women of childbearing potential must agree to use an effective method of birth control, as defined above, from enrolment, throughout the study duration and within the 8 treatment weeks. They must demonstrate a negative serum pregnancy test at screening and demonstrate a negative urine pregnancy test immediately before each dose of study drug or placebo. Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of randomization without an alternative medical cause. The following age-specific requirements apply:

    i. Women <50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.

    ii. Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
23. Male patients not using an acceptable method of contraception. All male patients who are sexually active must agree to use an acceptable method of contraception (condom with or without spermicide, vasectomy) from the first dose of study drug until their last dose.
24. Use of angiotensin-converting-enzyme inhibitors
25. Use of immunosuppressive medication (including but not limited to: methotrexate, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid, oral corticosteroid, or any experimental anti-inflammatory therapy) within 3 months prior to the date informed consent is obtained
26. Use of any other biological within 4 months or 5 half-lives prior to randomization, whichever is longer.
27. Any centrally acting medication within the last 2 weeks which in the view of the investigator could influence the coughing (Any participant who is taking amitriptyline, dextromethorphan, pregabalin, gabapentin or opioids will not be eligible to take part in this study unless they are willing and medically able to withdraw from such medication for the duration of the study. The reason for this is that centrally acting medications may influence coughing rates.)
28. History of psychiatric illness, drug or alcohol abuse which may interfere in the participation of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imran Satia, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schappert SM, Burt CW. Ambulatory care visits to physician offices, hospital outpatient departments, and emergency departments: United States, 2001-02. Vital Health Stat 13. 2006 Feb;(159):1-66. PMID 16471269
- [Background] Song WJ, Chang YS, Faruqi S, Kim JY, Kang MG, Kim S, Jo EJ, Kim MH, Plevkova J, Park HW, Cho SH, Morice AH. The global epidemiology of chronic cough in adults: a systematic review and meta-analysis. Eur Respir J. 2015 May;45(5):1479-81. doi: 10.1183/09031936.00218714. Epub 2015 Feb 5. No abstract available. PMID 25657027
- [Background] Irwin RS, Baumann MH, Bolser DC, Boulet LP, Braman SS, Brightling CE, Brown KK, Canning BJ, Chang AB, Dicpinigaitis PV, Eccles R, Glomb WB, Goldstein LB, Graham LM, Hargreave FE, Kvale PA, Lewis SZ, McCool FD, McCrory DC, Prakash UBS, Pratter MR, Rosen MJ, Schulman E, Shannon JJ, Hammond CS, Tarlo SM. Diagnosis and management of cough executive summary: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):1S-23S. doi: 10.1378/chest.129.1_suppl.1S. No abstract available. PMID 16428686
- [Background] French CL, Irwin RS, Curley FJ, Krikorian CJ. Impact of chronic cough on quality of life. Arch Intern Med. 1998 Aug 10-24;158(15):1657-61. doi: 10.1001/archinte.158.15.1657. PMID 9701100
- [Background] Brightling CE, Ward R, Goh KL, Wardlaw AJ, Pavord ID. Eosinophilic bronchitis is an important cause of chronic cough. Am J Respir Crit Care Med. 1999 Aug;160(2):406-10. doi: 10.1164/ajrccm.160.2.9810100. PMID 10430705
- [Background] Gibson PG, Dolovich J, Denburg J, Ramsdale EH, Hargreave FE. Chronic cough: eosinophilic bronchitis without asthma. Lancet. 1989 Jun 17;1(8651):1346-8. doi: 10.1016/s0140-6736(89)92801-8. PMID 2567371
- [Background] Carney IK, Gibson PG, Murree-Allen K, Saltos N, Olson LG, Hensley MJ. A systematic evaluation of mechanisms in chronic cough. Am J Respir Crit Care Med. 1997 Jul;156(1):211-6. doi: 10.1164/ajrccm.156.1.9605044. PMID 9230750
- [Background] Satia I, Watson R, Scime T, Dockry RJ, Sen S, Ford JW, Mitchell PD, Fowler SJ, Gauvreau GM, O'Byrne PM, Smith JA. Allergen challenge increases capsaicin-evoked cough responses in patients with allergic asthma. J Allergy Clin Immunol. 2019 Sep;144(3):788-795.e1. doi: 10.1016/j.jaci.2018.11.050. Epub 2019 Jan 17. PMID 30660644
- [Background] Drake MG, Scott GD, Blum ED, Lebold KM, Nie Z, Lee JJ, Fryer AD, Costello RW, Jacoby DB. Eosinophils increase airway sensory nerve density in mice and in human asthma. Sci Transl Med. 2018 Sep 5;10(457):eaar8477. doi: 10.1126/scitranslmed.aar8477. PMID 30185653
- [Derived] Diab N, Brister D, Kum E, Wahab M, Hassan W, Beaudin S, Obminski C, Wattie J, Wiltshire L, Howie K, Killian K, Holt K, Sehmi R, Gauvreau GM, Smith JA, O'Byrne PM, Satia I. Mepolizumab for the treatment of refractory chronic cough in patients with eosinophilic airways disease (MUCOSA): a randomized, double-blind, parallel-group, placebo-controlled trial. Eur Respir J. 2025 Nov 6:2501573. doi: 10.1183/13993003.01573-2025. Online ahead of print. PMID 41198391

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Arm: Normal Saline (0.9% normal saline) Dosage form: 1ml pre-filled syringe Dosage: n/a Frequency: 4 doses at days 0, 28, 56 and 84 Duration: 12 weeks
  Normal Saline: Placebo subcutaneous injection administered 4 times days 0, 28, 56 and 84 during 12 week treatment period.
Period: Overall Study
Arm/Group | Mepolizumab Arm | Placebo Arm
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Mepolizumab Arm: Mepolizumab Dosage form: 1 ml pre-filled syringe Dosage: 100 mg Frequency: 4 doses at days 0, 28, 56 and 84 Duration: 12 weeks
  Mepolizumab: Mepolizumab subcutaneous injection administered 4 times days 0, 28, 56 and 84 during 12 week treatment period.
- Total: Total of all reporting groups
Arm/Group | Mepolizumab Arm | Placebo Arm | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.87 (9.72) | 65.80 (13.93) | 65.83 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 13 | 14 | 27
  Race/Ethnicity: Other | 2 | 1 | 3
Region of Enrollment [Number; unit: Participants]
  Canada | 15 | 15 | 30
Cough Duration (months) [Median (Full Range); unit: Months] | 120 [25 to 588] | 61 [11 to 228] | 115.5 [11 to 588]
Diagnosis [Count of Participants; unit: Participants]
  Non-asthmatic eosinophilic bronchitis | 7 | 4 | 11
  Asthma | 8 | 11 | 19
% Sputum Eosinophils [Median (Full Range); unit: Percentage] | 2.6 [2.0 to 11.8] | 2.6 [2.0 to 6.2] | 2.6 [2.0 to 11.8]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Cough Frequency at 14 Weeks
Description: Change from baseline in 24-hour cough frequency (coughs/hour) measured by the VitaloJAK cough monitor at 14 weeks.
Time Frame: 14 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
Coughs/hour
  Week 0 | 17.0 [16.7 to 17.3] | 17.0 [16.7 to 17.3]
  Week 14 | 12.6 [8.2 to 19.3] | 10.6 [7.6 to 15.0]
Statistical Analysis 1: Comparison: Mepolizumab Arm vs Placebo Arm; The primary outcome was the change from baseline in log-transformed 24-hour cough frequency (coughs/hour) at week 14; Test type: Superiority; p = 0.99, Generalized estimating equations — The model included treatment group, week, the interaction between treatment group and week, and baseline log-transformed 24-hour cough frequency as fixed effects; Hypothesis tests were two-sided, a p<0.05 indicated statistical significance. We made no adjustments for multiple comparisons across outcomes; % change relative to placebo = 18, 95% CI 2-sided [-46.4 to 160.1]

2. Secondary Outcome: Change From Baseline in Awake Cough Frequency at 8 Weeks
Description: Change from baseline in awake cough frequency (coughs/hour) measured by the VitaloJAK cough monitor at 8 weeks.
Time Frame: 8 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
Coughs/hour
  Week 0 | 22.5 [22.4 to 22.6] | 22.5 [22.5 to 22.6]
  Week 8 | 17.8 [13.8 to 23.0] | 12.5 [10.8 to 14.6]

3. Secondary Outcome: Change From Baseline in Awake Cough Frequency at 14 Weeks
Description: Change from baseline in awake cough frequency (coughs/hour) at 14 weeks.
Time Frame: 14 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
Coughs/hour
  Week 0 | 22.5 [22.4 to 22.6] | 22.5 [22.5 to 22.6]
  Week 14 | 16.3 [10.6 to 25.1] | 14.1 [9.7 to 20.4]

4. Secondary Outcome: Change From Baseline in Sleep Cough Frequency at 8 Weeks
Description: Change from baseline in sleep cough frequency (coughs/hour) measured by the VitaloJAK cough monitor at 8 weeks.
Time Frame: 8 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
Coughs/hour
  Week 0 | 1.8 [1.5 to 2.3] | 1.7 [1.3 to 2.2]
  Week 8 | 1.0 [0.5 to 2.1] | 1.4 [0.7 to 2.8]

5. Secondary Outcome: Change From Baseline in Sleep Cough Frequency at 14 Weeks
Description: Change from baseline in sleep cough frequency (coughs/hour) measured by the VitaloJAK cough monitor at 14 weeks.
Time Frame: 14 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
Coughs/hour
  Week 0 | 1.8 [1.5 to 2.3] | 1.7 [1.3 to 2.2]
  Week 14 | 1.9 [0.9 to 4.0] | 1.5 [0.9 to 2.4]

6. Secondary Outcome: Change From Baseline in Cough Severity at 8 Weeks
Description: Change from baseline in cough severity measured on the 100-mm visual analogue scale at 8 weeks. Scale ranges from 0 mm (no cough) to 100 mm (worst possible cough). Higher scores reflect worse cough severity.
Time Frame: 8 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
mm
  Week 0 | 65.3 [62.1 to 68.5] | 63.9 [60.7 to 67.0]
  Week 8 | 55.7 [45.4 to 66.0] | 49.3 [41.9 to 56.8]

7. Secondary Outcome: Change From Baseline in Cough Severity at 14 Weeks
Description: Change from baseline in cough severity measured on the 100-mm visual analogue scale at 14 weeks. Scale ranges from 0 mm (no cough) to 100 mm (worst possible cough). Higher scores reflect worse cough severity.
Time Frame: 14 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
mm
  Week 0 | 65.3 [62.1 to 68.5] | 63.9 [60.7 to 67.0]
  Week 14 | 49.5 [35.9 to 63.1] | 51.4 [40.8 to 62.0]

8. Secondary Outcome: Change From Baseline on the Leicester Cough Questionnaire at 8 Weeks
Description: Change from baseline in cough quality of life measured by the Leicester Cough Questionnaire at 8 weeks. Total score ranges from 3 to 21, with higher scores indicating better cough quality of life.
Time Frame: 8 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
points
  Week 0 | 11.3 [10.8 to 11.8] | 11.1 [10.5 to 11.6]
  Week 8 | 11.6 [10.0 to 13.2] | 13.7 [12.4 to 14.9]

9. Secondary Outcome: Change From Baseline on the Leicester Cough Questionnaire at 14 Weeks
Description: Change from baseline in cough quality of life measured by the Leicester Cough Questionnaire at 14 weeks. Total score ranges from 3 to 21, with higher scores indicating better cough quality of life.
Time Frame: 14 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
points
  Week 0 | 11.3 [10.8 to 11.8] | 11.1 [10.5 to 11.6]
  Week 14 | 12.8 [11.1 to 14.6] | 13.7 [12.3 to 15.0]

10. Secondary Outcome: Change From Baseline in Blood Eosinophils at 8 Weeks
Description: Change from baseline in blood eosinophils at 8 weeks.
Time Frame: 8 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Mean (95% Confidence Interval); unit: cells/µL
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
cells/µL
  Week 0 | 284.2 [256.1 to 312.2] | 288.9 [259.1 to 318.8]
  Week 8 | 57.5 [19.4 to 95.6] | 282.2 [191.0 to 373.6]

11. Secondary Outcome: Change From Baseline in Blood Eosinophils at 14 Weeks
Description: Change from baseline in blood eosinophils at 14 weeks.
Time Frame: 14 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Mean (95% Confidence Interval); unit: cells/µL
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
cells/µL
  Week 0 | 284.2 [256.1 to 312.2] | 288.9 [259.1 to 318.8]
  Week 14 | 44.2 [4.0 to 84.3] | 281.9 [242.9 to 320.9]

12. Secondary Outcome: Change From Baseline in Sputum Eosinophils at 8 Weeks
Description: Change from baseline in sputum eosinophils (%) at 8 weeks.
Time Frame: 8 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: % sputum eosinophils
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
% sputum eosinophils
  Week 0 | 2.9 [2.4 to 3.4] | 2.8 [2.4 to 3.2]
  Week 8 | 1.8 [1.3 to 2.6] | 2.8 [2.0 to 3.8]

13. Secondary Outcome: Change From Baseline in Sputum Eosinophils at 14 Weeks
Description: Change from baseline in sputum eosinophils (%) at 14 weeks.
Time Frame: 14 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: % sputum eosinophils
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
% sputum eosinophils
  Week 0 | 2.9 [2.4 to 3.4] | 2.8 [2.4 to 3.2]
  Week 14 | 1.6 [1.0 to 2.4] | 2.6 [1.7 to 4.1]

14. Other Pre Specified Outcome: Change From Baseline in Methacholine Provocative Concentration Eliciting a 20% Fall in FEV1 (PC20) at 14 Weeks
Description: Change from baseline in methacholine provocative concentration eliciting a 20% fall in FEV1 (PC20) at 14 weeks.
Time Frame: 14 weeks
Population: All patients who received at least one dose of a study drug were included in a modified intention-to-treat analysis.
Measure: Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | Mepolizumab Arm | Placebo Arm
Number analyzed (Participants) | 15 | 15
mg/mL
  Week -2 | 14.4 [12.4 to 16.4] | 13.1 [11.1 to 15.1]
  Week 14 | 15.8 [9.1 to 22.5] | 24.3 [19.1 to 29.5]

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: All adverse events were reported.
Arm/Group | Mepolizumab Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab Arm (N=15) | Placebo Arm (N=15)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT04765722/Prot_SAP_000.pdf